CLINICAL TRIAL: NCT02644070
Title: A Prospective Randomized-controlled Multicenter Clinical and Histological Study of Extraction Site Augmentation With mp3 vs. Apatos
Brief Title: mp3 vs Apatos in Post-extractive Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuscan Dental Institute (Other)
Responsible Party: Principal Investigator, Antonio Barone, Antonio Barone, DDS, PhD, MSc, University of Pisa Adjunct Professor, Tuscan Dental Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 214 in June 14, 2012
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Alveolar Bone Loss
Keywords: Alveolar bone loss; Alveoloplasty; Bone remodeling; Xenograft; Tooth socket; Dental implant
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- alveolar bone preservation with mp3 (Experimental): Extraction sockets grafted with corticocancellous porcine bone and collagen (MP3, Osteobiol, Coazze, Italy) with graft particle size between 600 and 1000 µm and a collagen membrane (Evolution, Osteobiol, Coazze, Italy) used to stabilize the biomaterial into the socket.
  Interventions: Device: alveolar bone preservation with mp3; Device: stabilization with membrane
- alveolar bone preservation with apatos (Experimental): Extraction sockets grafted with cortical porcine bone with particle size between 600 and 1000 µm (Apatos, Osteobiol, Coazze, Italy ) and a collagen membrane (Evolution, Osteobiol, Coazze, Italy) used to stabilize the biomaterial into the socket.
  Interventions: Device: alveolar bone preservation with apatos; Device: stabilization with membrane
- NO_graft (No Intervention): extraction sockets with spontaneous healing

INTERVENTIONS:
Device: alveolar bone preservation with mp3 — graft with corticocancellous porcine bone and collagen (MP3, Osteobiol, Coazze, Italy)
  Arms: alveolar bone preservation with mp3
Device: alveolar bone preservation with apatos — graft with cortical porcine bone (Apatos, Osteobiol, Coazze, Italy )
  Arms: alveolar bone preservation with apatos
Device: stabilization with membrane — socket stabilization with a collagen membrane (Evolution, Osteobiol, Coazze, Italy)
  Arms: alveolar bone preservation with apatos; alveolar bone preservation with mp3

SUMMARY:
The primary aim of the present multicenter randomized controlled trial was to evaluate and compare the shortterm clinical and histological changes of extraction sockets after ridge preservation procedures with changes of extraction sockets that healed naturally.

The secondary aim was to evaluate which, if any extraction socket characteristics could have affected tissue changes occurring at the augmented as well as naturally healed sites.

Recruitment and enrollment of patients were performed from June 2011 to June 2012 in five university centers/private practice:

* University of Pisa;
* University of Murcia;
* University of Ancona;
* Private practice, Dr. Di Felice;
* University of Verona.

Randomization:

1. extraction sockets with spontaneous healing;
2. extraction sockets grafted with pre-hydrated collagenated cortico-cancellous porcine bone, with a particle size between 600 and 1000 μm;
3. extraction sockets grafted with cortical porcine bone, with a particle size between 600 and 1000 μm.

Outcome Variables

* Complications
* Changes of ridge volume contour;
* Vertical bone changes;
* Buccal-Lingual Width;
* Histomorphometric parameters.

Sample size was calculated comparing outcome data between grafted sockets versus non-grafted sockets. The primary parameter was the change in mid-buccal vertical height (0.7±1.4mm and 3.6±1.5mm, respectively, for the test and control groups) (Barone et al. 2008). Final sample size was increased to 30 subjects per group due to possible patient dropout events. Each center contributed according to the predetermined 1:1:1 ratio; the fresh extraction socket was considered the unit of randomization.

Corrections for balancing the three experimental groups for confounding factors were not applied.

A matrix elaborator performed all the analyses§§: multi-way analysis of variance (ANOVAn) was applied, then appropriate post hoc comparison tests were run; post hoc estimated effect sizes were calculated with a power of 0.9. The level of statistical significance was set at 0.05 for all analyses.

DETAILED DESCRIPTION:
BACKGROUND

Following tooth extraction, the alveolar ridge undergoes a marked change. During the first year after tooth extraction, about 50% of the bucco-lingual ridge dimension will be lost. Furthermore, ridge reduction will become more pronounced from a buccal than from a lingual/palatal aspect. The hard tissue modelling and remodelling following tooth extraction were studied in the dog model. It was demonstrated that the socket was first occupied by a coagulum that was replaced with granulation tissue, provisional connective tissue and woven bone. This immature hard tissue was subsequently replaced with lamellar bone and bone marrow. During the healing phase, the height of the buccal bone wall was substantially reduced. In addition, about 30% of the marginal portion of the alveolar process of the extraction site was lost.

Several approaches have been tested to preserve or improve the dimension and contour of the ridge following tooth extraction including the use of various graft or filler materials such as autografts, allografts, xenografts and/ or barrier membranes. The most recent studies on animals as well as in humans showed that the placement of xenografts in fresh extraction sockets promoted de novo hard tissue formation, in particular in the marginal portion of the extraction site. Moreover, it should be considered that the dimension of hard tissue walls was maintained and the profile of the ridge preserved. The data concerning socket preservation techniques in humans are still scarce. Therefore, firm conclusions about dimensional changes cannot be drawn currently; in reality, socket preservation procedures may aid in reducing the bone dimensional changes following tooth extraction. However, they do not completely prevent bone resorption so that a loss in width and height may be still expected; even if this procedure can allows a better location for implant placement and minimize the need for GBR procedure simultaneously with implant placement when compared to natural healed sites.

The histologic and histomorphometric evaluations showed the early phase of hard tissue formation were altered in extraction sockets that were grafted with a deproteinized bovine bone mineral immediately after tooth removal. The authors suggested that this modified wound healing and bone modelling may have been influenced by the presence of multinucleated cells that occurred in tissues harbouring the xenogenic graft. Thus, in grafted sites, substantial amount of newly formed bone could only be detected in the apical portion of the sockets where the graft material was absent. In the remaining portions of the grafted sockets a mildly inflamed provisional matrix surrounded the majority of bovine bone mineral particles, whose surface was frequently, but not always, coated with multinucleated cells. The biological behaviour can be explained with the type of biomaterial which is not resorbable/or slowly resorbable.

Given these premises, this prospective, randomized-controlled multicenter clinical study will compare the dimensional healing pattern, the quality of de novo bone formation and the implant placement in large tooth extraction sites after grafting with two types of xenografts: MP3 vs. Apatos by Tecnoss- Osteobiol.

Specific objectives:

* To augment fresh premolar and molar extraction sites with MP3 and Apatos;
* To evaluate dimensional ridge changes with MP3 and Apatos ( clinical measurements and volumetric evaluations with a computerized analysis of study casts);
* To place implants (BT EVO, Biotec, Povolaro, Italy) 3 months after grafting ( diameter, length, need for additional GBR procedures);
* To evaluate the histological aspects of bone biopsies taken at the osteotomy preparation sites;
* To follow and to monitor the implant success in treated sites for up to 24 months.

The present study tested as first outcome the null hypothesis that there were no differences between the 2 biomaterials against the alternative hypothesis of a difference;

- second long-term outcome performance of implants placed in grafted sites. .

Statistical Analysis The sample size was calculated for the primary outcome measures (implant failure); it was decided to recruit 30 patients in each group.

Data analysis was performed with descriptive statistics and independent sample t-test was used for comparison of mean values between groups to evaluate the significant differences between the two treatment groups. The Pearson Chi Square test was used to test for relationships between variables. A p value <0.05 was selected as the level of statistical significance. The estimation of the implant survival rate was based on Kaplan-Meier analysis. Cumulative implant survival over time was assessed using the Kaplan-Meyer analysis. The cumulative survival rate (CSR) is the probability that the implant will survive at least to a stated time within the observation period of the investigation. The failure time for each implant was defined as the elapsed time from placement to the date of failure. In cases where the terminal event was not reached, the elapsed time between implant insertion and last visit was assumed as the survival time. All evaluations were performed using SPSS software version 6.1.2 for Windows.

STUDY PROCEDURES

Visit 1 Pre-surgical assessment Patients will be seen for evaluation and enrolment. Upon enrolment an informed consent form will be signed by the patient prior to enrolment in the study after which a patient study number will be assigned. Documentation of demographic, medical and dental conditions and pre-operative site conditions will be recorded on a specific case report form. Impressions will be taken to obtain an individualized template which will be used for clinical measurements after tooth extraction.

VISIT 2 Tooth Extraction and Grafting Procedure All surgeries have to be performed with the same technique by calibrated clinicians. After dental extraction, the resulting sockets will be debrided and clinical measurements evaluated. The number of extracted tooth will be recorded on a specific case report form. Impressions will be taken to obtain study casts to evaluate volumetric changes of the extraction socket site with the use of a computerized software system.

At completion of tooth extraction efforts, the patient's randomization card will be unmasked to reveal the treatment group assignment for each extraction site.

For the purpose of this study it will be necessary to ensure the removal of all remaining root fragments, fibers and soft tissue from the sockets prior to placement of graft material. Either curettes and/or burs may be used for degranulation of extraction sockets. The following extraction procedure observations will be documented: methods used for tooth removal, need for curettage of extraction site.

Each alveolar socket will be classified according the following classification in addition [ Joudzbalys et al. 2008 and 2010].

Type Classification Type I Socket The facial soft tissue an buccal plate of bone are at normal levels in relation to the cementoenamel junction of the pre-extracted tooth and remain intact postextraction Type II Socket Facial soft tissue is present but the buccal plate is partially missing following extraction of the tooth.

Type III Socket The facial soft tissue and the buccal plate of bone are both markedly reduced after tooth extraction.

Grafting material will handled according to manufacturer's recommendations and each extraction site will receive the graft type that has been assigned according to randomization scheme. Do not over compact. The patient's blood is the preferred hydration material for mixing with the graft material.

The use of a collagen membrane is mandatory in order to ensure capture of the graft material. The Evolution membrane will be trimmed according the size of the defect and will be adapted over the bone cavity in attaching the ends underneath the adjacent soft tissue. The mucosal margins will be fixed in place in using "mattress sutures". Removal of sutures will take place ten (10) days thereafter. Information on all surgical materials used in the alveolar socket procedures that remain in the patient and any other ancillary procedures used to treat the patient will be documented in the according Case Report Form.

Post surgical medications should be standardized for all study patients, see the above reported material and methods section.

Photographs of each of the treated sites will be done to document the condition of the site.

Preparation of a bite blocks are essential to ensure proper radiographic alignment for subsequent periapical radiographs ( see materials and methods section). A periapical radiograph will be obtained for each study alveolar socket after tooth extraction to determine if complete removal of the teeth has been achieved. Please provide the radiographic files with the patient study identification, the date, and the tooth site number. For centers using conventional radiographic films, only original radiographs can be used for evaluation and analysis. The use of duplicate original film will therefore be needed.

VISIT 3 Healing Assessment (10 days)

Patients will return to clinic and be examined for healing assessment and suture removal. Patients will be interviewed for determination of any signs or symptoms of medical events. Clinical assessments of the treated sites will be done as described in the Special Procedures section. The condition of the membrane will be documented. After suture removal the sites will be inspected to ensure the proper seating of the membrane and that no spillage of graft material is observed. All information will be documented on the specific Case Report Form.

Visit 4 Membrane Assessment (Month 1)

The patients will return for membrane healing assessment. The condition of the membrane will be documented and registered.

Impressions will be taken to obtain study casts to evaluate volumetric changes of the extraction socket site with the use of a computerized software system.

Visit 5 Implant Placement ( Month 4 )

An evaluation of the implant sites will be done prior to the implant placement procedures. If any residues of the collagen membrane will be observed the findings will be documented.

Impressions will be taken to obtain study casts to evaluate volumetric changes of the extraction socket site with the use of a computerized software system.

A perioprobe will be used to measure the thickness of the mucosa at the crestal center and the buccal (3 mm distant from central aspect) lingual position (3 mm distant from the central aspect) of where the implant will be placed. These values will be recorded in millimeters.

Mucoperiosteal flap has to be raised and clinical measurements were taken using an individualized template. All surgeries will be performed under clean conditions keeping the implant sterile throughout placement. Procedures indicated in Biotec surgical manual will be followed and final drilling should be performed with low speed, high torque, irrigating hand piece and drills.

As part of preparing the osteotomy site, a trephine drill will be used and all bone material removed with the drill will be preserved for histological analysis. The length of the core needs to be 6 to 8 mm to be sufficient for analysis.

The specific dimensions of the implant will be at the discretion of the investigator. The implant catalog and lot numbers will be documented. At completion of implant placement procedures record the ultimate position of the seating surface: Sup = supracrestal, Cres = crestal, or Sub = subcrestal. All information including the position and the size of the chosen implants will be documented on the appropriate Case Report Form. Moreover, the need for simultaneous GBR procedures should be registered.

The final torque and use of the ratchet will be recorded along with the amount of rotation applied to the implant on the appropriate Case Report Form.

A periapical radiograph will be obtained of all grafted sites (at the beginning of the visit) and an additional one will be taken of all study implants after the implant placement surgery is completed.

Visit 6 Healing Assessment( 1 Week Post-implant Placement)

An evaluation of the status of the implant surgical sites will be done. Scores for gingival inflammation, gingival and plaque indices, implant mobility, peri-implant radiolucency and suppuration will be recorded on appropriate Case Report Form. An evaluation of the patient's oral health will be done by scoring gingival and plaque indices as described in the Special Procedures section. The final restoration is at the discretion of the investigator and according to the treatment plan design within six (6) months of implant placement.

The insertion of a temporary prosthesis will be accomplished at the investigator's discretion; he may also fabricate the final restoration directly. The insertion of the restoration will not take place before four months in the mandible and six on the maxilla after implant placement surgery the delivery of the final prosthesis will be completed. Information on prosthesis composition, insertion, outcome, anchorage and abutments used will be recorded on the appropriate Case Report Form.

Visit 7, 8 and 9 Clinical Assessment (12, 18 and 24 Months)

Follow-up evaluations will be carried out at six month intervals following implant placement surgery for two years. At each follow-up interval, patients will return to the clinic for assessment of implant and periodontal tissue. A periapical radiograph of all study implants will be obtained. All data gathered at these evaluations will be recorded on appropriate Case Report Forms. Scores for site-specific gingival inflammation, gingival and plaque indices, implant mobility, peri-implant radiolucency, and suppuration will be recorded on appropriate Case Report Form. An evaluation of the patient's oral health will be done by scoring gingival and plaque indices as described in the Special Procedures section.

By the end of 6 months after implant placement surgery the delivery of the final prosthesis will be completed. Information on prosthesis composition, insertion, outcome, anchorage and abutments used will be recorded on appropriate Case Report Form.

PROTOCOL AMENDMENTS

Any proposed change to the protocol is to be discussed with the clinical monitor in a timely manner. Once both the investigators and the sponsor have accepted the changes by, a written addendum to the protocol or a revised protocol will be sent to the investigators for signature. Copies of addenda and revised protocols will be kept by both parties in their respective files.

PROTOCOL DEVIATIONS AND VIOLATIONS

Occasionally during the study, deviations from the procedures established in the protocol may occur. Any deviation from the protocol is reason to contact the clinical monitor without delay. The deviation will be documented on the Patient Status Form. Enrollment and treatment of patients who do not meet Admission Criteria will be considered a protocol violation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* requiring one single tooth extraction and subsequently an implant-supported restoration
* able to sign an informed consent form

Exclusion Criteria:

* history of systemic diseases that would contraindicate oral surgical treatment;
* long-term non-steroidal anti-inflammatory drug therapy;
* lack of opposite occluding dentition in the area intended for extraction and subsequent implant placement;
* Oral biphosphonate therapy;
* absence of adjacent teeth;
* unwillingness to return for the follow-up examination;
* use of more than 10 cigarettes per day. Subjects smoking less than 10 cigarettes per day were requested to stop smoking before and after surgery; however, their compliance could not be monitored.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Clinical vertical bone changes | 0 months after grafting
  Vertical bone changes were evaluated in mm with the use of a custom made stent at mesial, distal, buccal and lingual/palatal sites; it was set as the distance between the reference point and the most apical point of the marginal bone level. Changes at the vertical bone level were evaluated by subtracting the postoperative value from the respective baseline value.
Clinical vertical bone changes | 1 month after grafting
  Vertical bone changes were evaluated in mm with the use of a custom made stent at mesial, distal, buccal and lingual/palatal sites; it was set as the distance between the reference point and the most apical point of the marginal bone level. Changes at the vertical bone level were evaluated by subtracting the postoperative value from the respective baseline value.
Clinical vertical bone changes | 3 months after grafting
  Vertical bone changes were evaluated in mm with the use of a custom made stent at mesial, distal, buccal and lingual/palatal sites; it was set as the distance between the reference point and the most apical point of the marginal bone level. Changes at the vertical bone level were evaluated by subtracting the postoperative value from the respective baseline value.
Clinical vertical bone changes | 12 months after grafting
  Vertical bone changes were evaluated in mm with the use of a custom made stent at mesial, distal, buccal and lingual/palatal sites; it was set as the distance between the reference point and the most apical point of the marginal bone level. Changes at the vertical bone level were evaluated by subtracting the postoperative value from the respective baseline value.
Clinical vertical bone changes | 24 months after grafting
  Vertical bone changes were evaluated in mm with the use of a custom made stent at mesial, distal, buccal and lingual/palatal sites; it was set as the distance between the reference point and the most apical point of the marginal bone level. Changes at the vertical bone level were evaluated by subtracting the postoperative value from the respective baseline value.
Clinical vertical bone changes | 36 months after grafting
  Vertical bone changes were evaluated in mm with the use of a custom made stent at mesial, distal, buccal and lingual/palatal sites; it was set as the distance between the reference point and the most apical point of the marginal bone level. Changes at the vertical bone level were evaluated by subtracting the postoperative value from the respective baseline value.
Volume of the alveolar ridge | 0 months after grafting
  Several impressions of the experimental sites were obtained from each patient. Impressions of the jaw were obtained in a one-step process with two viscosity polyvinyl siloxane impression materials. Within 24 h, model casts of the dental impressions were obtained using plaster of Paris. A scanner for cone-beam computerized tomography was employed for 3D file acquisition of the different model casts of each patient. The CBCT scan data were inserted into a Matrix Laboratory, and for each patient, positions of axial images related to all time frames were elaborated in space in such a way that the residual teeth were superimposable (Sbordone et al. 2012a,b); A volumetric evaluation (V in cm3) of the study models in the site subjected to alveolar ridge preservation was performed with Segment and Planning tool of SimPlant Pro 12.02.
Volume of the alveolar ridge | 1 month after grafting
  Several impressions of the experimental sites were obtained from each patient. Impressions of the jaw were obtained in a one-step process with two viscosity polyvinyl siloxane impression materials. Within 24 h, model casts of the dental impressions were obtained using plaster of Paris. A scanner for cone-beam computerized tomography was employed for 3D file acquisition of the different model casts of each patient. The CBCT scan data were inserted into a Matrix Laboratory, and for each patient, positions of axial images related to all time frames were elaborated in space in such a way that the residual teeth were superimposable (Sbordone et al. 2012a,b); A volumetric evaluation (V in cm3) of the study models in the site subjected to alveolar ridge preservation was performed with Segment and Planning tool of SimPlant Pro 12.02.
Volume of the alveolar ridge | 3 months after grafting
  Several impressions of the experimental sites were obtained from each patient. Impressions of the jaw were obtained in a one-step process with two viscosity polyvinyl siloxane impression materials. Within 24 h, model casts of the dental impressions were obtained using plaster of Paris. A scanner for cone-beam computerized tomography was employed for 3D file acquisition of the different model casts of each patient. The CBCT scan data were inserted into a Matrix Laboratory, and for each patient, positions of axial images related to all time frames were elaborated in space in such a way that the residual teeth were superimposable (Sbordone et al. 2012a,b); A volumetric evaluation (V in cm3) of the study models in the site subjected to alveolar ridge preservation was performed with Segment and Planning tool of SimPlant Pro 12.02.
Volume of the alveolar ridge | 12 months after grafting
  Several impressions of the experimental sites were obtained from each patient. Impressions of the jaw were obtained in a one-step process with two viscosity polyvinyl siloxane impression materials. Within 24 h, model casts of the dental impressions were obtained using plaster of Paris. A scanner for cone-beam computerized tomography was employed for 3D file acquisition of the different model casts of each patient. The CBCT scan data were inserted into a Matrix Laboratory, and for each patient, positions of axial images related to all time frames were elaborated in space in such a way that the residual teeth were superimposable (Sbordone et al. 2012a,b); A volumetric evaluation (V in cm3) of the study models in the site subjected to alveolar ridge preservation was performed with Segment and Planning tool of SimPlant Pro 12.02.
Volume of the alveolar ridge | 24 months after grafting
  Several impressions of the experimental sites were obtained from each patient. Impressions of the jaw were obtained in a one-step process with two viscosity polyvinyl siloxane impression materials. Within 24 h, model casts of the dental impressions were obtained using plaster of Paris. A scanner for cone-beam computerized tomography was employed for 3D file acquisition of the different model casts of each patient. The CBCT scan data were inserted into a Matrix Laboratory, and for each patient, positions of axial images related to all time frames were elaborated in space in such a way that the residual teeth were superimposable (Sbordone et al. 2012a,b); A volumetric evaluation (V in cm3) of the study models in the site subjected to alveolar ridge preservation was performed with Segment and Planning tool of SimPlant Pro 12.02.
Volume of the alveolar ridge | 36 months after grafting
  Several impressions of the experimental sites were obtained from each patient. Impressions of the jaw were obtained in a one-step process with two viscosity polyvinyl siloxane impression materials. Within 24 h, model casts of the dental impressions were obtained using plaster of Paris. A scanner for cone-beam computerized tomography was employed for 3D file acquisition of the different model casts of each patient. The CBCT scan data were inserted into a Matrix Laboratory, and for each patient, positions of axial images related to all time frames were elaborated in space in such a way that the residual teeth were superimposable (Sbordone et al. 2012a,b); A volumetric evaluation (V in cm3) of the study models in the site subjected to alveolar ridge preservation was performed with Segment and Planning tool of SimPlant Pro 12.02.
Buccal-Lingual Width | 0 months after grafting
  Buccal-Lingual Width was evaluated in mm, measuring the distance between buccal and lingual/palatal plate with a periodontal probe. Changes at bucco-lingual width were calculated by subtracting the baseline value from the post-operative value.
Buccal-Lingual Width | 1 month after grafting
  Buccal-Lingual Width was evaluated in mm, measuring the distance between buccal and lingual/palatal plate with a periodontal probe. Changes at bucco-lingual width were calculated by subtracting the baseline value from the post-operative value.
Buccal-Lingual Width | 3 months after grafting
  Buccal-Lingual Width was evaluated in mm, measuring the distance between buccal and lingual/palatal plate with a periodontal probe. Changes at bucco-lingual width were calculated by subtracting the baseline value from the post-operative value.
Buccal-Lingual Width | 12 months after grafting
  Buccal-Lingual Width was evaluated in mm, measuring the distance between buccal and lingual/palatal plate with a periodontal probe. Changes at bucco-lingual width were calculated by subtracting the baseline value from the post-operative value.
Buccal-Lingual Width | 24 months after grafting
  Buccal-Lingual Width was evaluated in mm, measuring the distance between buccal and lingual/palatal plate with a periodontal probe. Changes at bucco-lingual width were calculated by subtracting the baseline value from the post-operative value.
Buccal-Lingual Width | 36 months after grafting
  Buccal-Lingual Width was evaluated in mm, measuring the distance between buccal and lingual/palatal plate with a periodontal probe. Changes at bucco-lingual width were calculated by subtracting the baseline value from the post-operative value.
Marginal bone loss | 12 months after grafting
  Bone loss was measured (in mm) by comparing the radiographs taken at baseline (immediately after placement) to the postoperative ones. The marginal bone height (MBL) was measured as the distance between the reference point (fixture-abutment interface) and the most apical point of the marginal bone level. Calibration was performed using the known thread-pitch distance of the implants (pitch = 1.0 mm), and fixture diameter and length.
Marginal bone loss | 24 months after grafting
  Bone loss was measured (in mm) by comparing the radiographs taken at baseline (immediately after placement) to the postoperative ones. The marginal bone height (MBL) was measured as the distance between the reference point (fixture-abutment interface) and the most apical point of the marginal bone level. Calibration was performed using the known thread-pitch distance of the implants (pitch = 1.0 mm), and fixture diameter and length.
Marginal bone loss | 36 months after grafting
  Bone loss was measured (in mm) by comparing the radiographs taken at baseline (immediately after placement) to the postoperative ones. The marginal bone height (MBL) was measured as the distance between the reference point (fixture-abutment interface) and the most apical point of the marginal bone level. Calibration was performed using the known thread-pitch distance of the implants (pitch = 1.0 mm), and fixture diameter and length.
Implant success | 12, 24, 36 months after grafting
  Implant failure (count) was defined as implant mobility, removal of implants caused by progressive bone loss or infection. The stability of each implant was evaluated at the delivery of prosthetic restoration and 1 year after implant insertion and two metallic handles of dental instruments were used to evaluate the stability of single crowns. Success rates (in percentage) were calculated according to the criteria suggested by Buser and colleagues.
Implant success | 24 months after grafting
  Implant failure (count) was defined as implant mobility, removal of implants caused by progressive bone loss or infection. The stability of each implant was evaluated at the delivery of prosthetic restoration and 1 year after implant insertion and two metallic handles of dental instruments were used to evaluate the stability of single crowns. Success rates (in percentage) were calculated according to the criteria suggested by Buser and colleagues.
Implant success | 36 months after grafting
  Implant failure (count) was defined as implant mobility, removal of implants caused by progressive bone loss or infection. The stability of each implant was evaluated at the delivery of prosthetic restoration and 1 year after implant insertion and two metallic handles of dental instruments were used to evaluate the stability of single crowns. Success rates (in percentage) were calculated according to the criteria suggested by Buser and colleagues.

SECONDARY OUTCOMES:
NFB: newly formed bone | 3 months after extraction procedure
  Specimens were decalcified in ethylenediaminetetraacetic acid (10%) for a period of 2 weeks. Specimens were again X-rayed in order to verify the decalcification procedure. After dehydratation in graded series of ethanol, the specimens were embedded in paraffin, sectioned (3-5 μm sections), and stained with hematoxyline-eosine and modified Mallory aniline blue. Examinations were performed in a Nikon Eclipse 80i microscope≠≠ using X1.0 to X40 objectives for descriptive evaluation and morphometrical measurements. Histomorphometric measurements were performed in order to calculate the percentages (i.e., area fraction in %) of mineralized bone 3 months after extraction procedure. All measurements were determined by using an Easy image 2000 system≠≠ for area measurements. A mean value from 3 different areas was calculated giving percentages of the above.
RGP: residual graft particle | 3 months after extraction procedure
  Specimens were decalcified in ethylenediaminetetraacetic acid (10%) for a period of 2 weeks. Specimens were again X-rayed in order to verify the decalcification procedure. After dehydratation in graded series of ethanol, the specimens were embedded in paraffin, sectioned (3-5 μm sections), and stained with hematoxyline-eosine and modified Mallory aniline blue. Examinations were performed in a Nikon Eclipse 80i microscope≠≠ using X1.0 to X40 objectives for descriptive evaluation and morphometrical measurements. Histomorphometric measurements were performed in order to calculate the percentages (i.e., area fraction in %) of residual graft materials 3 months after extraction procedure. All measurements were determined by using an Easy image 2000 system≠≠ for area measurements. A mean value from 3 different areas was calculated giving percentages of the above.
NMT: non-mineralized tissue | 3 months after extraction procedure
  Specimens were decalcified in ethylenediaminetetraacetic acid (10%) for a period of 2 weeks. Specimens were again X-rayed in order to verify the decalcification procedure. After dehydratation in graded series of ethanol, the specimens were embedded in paraffin, sectioned (3-5 μm sections), and stained with hematoxyline-eosine and modified Mallory aniline blue. Examinations were performed in a Nikon Eclipse 80i microscope≠≠ using X1.0 to X40 objectives for descriptive evaluation and morphometrical measurements. Histomorphometric measurements were performed in order to calculate the percentages (i.e., area fraction in %) of non-mineralized tissue (i.e., connective tissue and/or bone marrow) 3 months after extraction procedure. All measurements were determined by using an Easy image 2000 system≠≠ for area measurements. A mean value from 3 different areas was calculated giving percentages of the above.
Facial Soft Tissue Level | 12 months after grafting
  Facial soft tissue levels (FST in mm) were evaluated, measuring the distance between level of soft tissues at mid-facial gingival level and a reference line, which connected the facial soft tissue level of the adjacent teeth. Facial soft tissue changes were calculated by subtracting the baseline value from the respective post-operative values according to the formula ΔFST = FST - FSTBaseline.
Facial Soft Tissue Level | 24 months after grafting
  Facial soft tissue levels (FST in mm) were evaluated, measuring the distance between level of soft tissues at mid-facial gingival level and a reference line, which connected the facial soft tissue level of the adjacent teeth. Facial soft tissue changes were calculated by subtracting the baseline value from the respective post-operative values according to the formula ΔFST = FST - FSTBaseline.
Facial Soft Tissue Level | 36 months after grafting
  Facial soft tissue levels (FST in mm) were evaluated, measuring the distance between level of soft tissues at mid-facial gingival level and a reference line, which connected the facial soft tissue level of the adjacent teeth. Facial soft tissue changes were calculated by subtracting the baseline value from the respective post-operative values according to the formula ΔFST = FST - FSTBaseline.
Width of keratinized gingiva | 12 months after grafting
  Width of keratinized gingiva (WKG in mm) was measured midfacially from the top of the edentulous crest to the mucogingival junction of the edentulous area before implant placement, and from the gingival margin to the mucogingival junction of the implanted site (after implant placement).
Width of keratinized gingiva | 24 months after grafting
  Width of keratinized gingiva (WKG in mm) was measured midfacially from the top of the edentulous crest to the mucogingival junction of the edentulous area before implant placement, and from the gingival margin to the mucogingival junction of the implanted site (after implant placement).
Width of keratinized gingiva | 36 months after grafting
  Width of keratinized gingiva (WKG in mm) was measured midfacially from the top of the edentulous crest to the mucogingival junction of the edentulous area before implant placement, and from the gingival margin to the mucogingival junction of the implanted site (after implant placement).
Papillae index | 12 months after grafting
  The status of the interdental papilla was recorded based on the index proposed by Jemt: 0 = no papilla; 1 = less than half the normal papilla height is present; 2 = greater than half the normal papilla height is present, but papilla does not extend to the normal contact point; 3 = papilla fills the entire proximal space and is in good harmony; 4 = papilla is hyperplastic.
Papillae index | 24 months after grafting
  The status of the interdental papilla was recorded based on the index proposed by Jemt: 0 = no papilla; 1 = less than half the normal papilla height is present; 2 = greater than half the normal papilla height is present, but papilla does not extend to the normal contact point; 3 = papilla fills the entire proximal space and is in good harmony; 4 = papilla is hyperplastic.
Papillae index | 36 months after grafting
  The status of the interdental papilla was recorded based on the index proposed by Jemt: 0 = no papilla; 1 = less than half the normal papilla height is present; 2 = greater than half the normal papilla height is present, but papilla does not extend to the normal contact point; 3 = papilla fills the entire proximal space and is in good harmony; 4 = papilla is hyperplastic.
Pink Esthetic Score | 12 months after grafting
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture . Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
  The mesial and distal papilla were evaluated for completeness, incompleteness or absence. All other variables were assessed by comparison with a reference tooth, i.e. the corresponding tooth (anterior region) or a neighboring tooth (premolar region).
Pink Esthetic Score | 24 months after grafting
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture . Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
  The mesial and distal papilla were evaluated for completeness, incompleteness or absence. All other variables were assessed by comparison with a reference tooth, i.e. the corresponding tooth (anterior region) or a neighboring tooth (premolar region).
Pink Esthetic Score | 36 months after grafting
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture . Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
  The mesial and distal papilla were evaluated for completeness, incompleteness or absence. All other variables were assessed by comparison with a reference tooth, i.e. the corresponding tooth (anterior region) or a neighboring tooth (premolar region).

REFERENCES:
- [Background] Barone A, Borgia V, Covani U, Ricci M, Piattelli A, Iezzi G. Flap versus flapless procedure for ridge preservation in alveolar extraction sockets: a histological evaluation in a randomized clinical trial. Clin Oral Implants Res. 2015 Jul;26(7):806-13. doi: 10.1111/clr.12358. Epub 2014 Mar 1. PMID 24580835
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Background] Barone A, Ricci M, Tonelli P, Santini S, Covani U. Tissue changes of extraction sockets in humans: a comparison of spontaneous healing vs. ridge preservation with secondary soft tissue healing. Clin Oral Implants Res. 2013 Nov;24(11):1231-7. doi: 10.1111/j.1600-0501.2012.02535.x. Epub 2012 Jul 12. PMID 22784417
- [Background] Covani U, Ricci M, Bozzolo G, Mangano F, Zini A, Barone A. Analysis of the pattern of the alveolar ridge remodelling following single tooth extraction. Clin Oral Implants Res. 2011 Aug;22(8):820-5. doi: 10.1111/j.1600-0501.2010.02060.x. Epub 2010 Dec 29. PMID 21198897
- [Background] Engler-Hamm D, Cheung WS, Yen A, Stark PC, Griffin T. Ridge preservation using a composite bone graft and a bioabsorbable membrane with and without primary wound closure: a comparative clinical trial. J Periodontol. 2011 Mar;82(3):377-87. doi: 10.1902/jop.2010.090342. Epub 2010 Nov 2. PMID 21043792
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475